CLINICAL TRIAL: NCT01210430
Title: Local Vasoconstriction in Postural Tachycardia Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Julian Stewart, Professor of Pediatrics, New York Medical College
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2R01HL074873-06A2 (NIH)
Record Dates: First submitted 2010-08-19; First posted 2010-09-28 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Postural Tachycardia Syndrome
Keywords: Postural Tachycardia Syndrome; Orthostatic Intolerance; Reactive Oxygen Species; Oxidative Stress; Angiotensin II; Nitric Oxide; Blood Flow; POTS; Ascorbic Acid; Vitamin C; Losartan
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance | interventions — Losartan; Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Losartan (Active Comparator)
  Interventions: Drug: Losartan
- Ascorbic Acid (VItamin C) (Active Comparator)
  Interventions: Drug: Ascorbic Acid (Vitamin C)
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Losartan — Subjects will receive placebo or losartan for 4 weeks. Days 1-7, subjects will receive 12.5mg of Losartan or placebo. Days 7-14, subjects will receive 25mg of Losartan or placebo. Days 14-28, subjects will receive 50mg of Losartan or placebo.
  Arms: Losartan
Drug: Ascorbic Acid (Vitamin C) — Subjects will receive 60mg/kg of Ascorbic Acid over 20 minutes followed by a maintenance infusion of 20mg/kg.
  Other Names: Vitamin C
  Arms: Ascorbic Acid (VItamin C)
Drug: Normal Saline — Subjects will receive 60mg/kg of normal saline over 20 minutes followed by a maintenance infusion of 20mg/kg of normal saline.
  Arms: Normal Saline

SUMMARY:
The investigators study will determine how often blood flow regulation abnormalities and abnormalities of sympathetic regulation produced by nitric oxide, angiotensin-II, and oxidative stress occur in POTS and the mechanism(s) of POTS in individual patients. Specific causes for POTS may vary from patient to patient. Patients will be compared to healthy control subjects. There is a treatment arm with a medication (losartan) that reduces the binding of angiotensin and increases NO. If the investigators know the specific biochemical mechanism the investigators may be able to offer further specific treatments to specific patients.

DETAILED DESCRIPTION:
Chronic orthostatic intolerance due to the postural tachycardia syndrome (POTS) severely impairs daily life in over a million Americans, mostly young women. POTS is defined by symptoms of orthostatic intolerance associated with excessive upright heart rate. While there is general agreement that abnormalities in vascular regulation and autonomic activity account for the tachycardia and symptoms of POTS, its pathophysiology is heterogeneous and only partially characterized.

The key feature of POTS is symptoms which are most prominent when standing. However, in some, findings are present supine (lying down) but worsened standing. Symptoms of POTS include dizziness in all patients, exercise provoked symptoms and thus exercise intolerance, excessive fatigue, nausea and abdominal pain, headache, shortness of breath and deep breathing, weakness, shakiness and postural anxiety, pallor, and neurocognitive loss (difficulty thinking). These occur on a day-to-day basis. The symptoms overlap with the case definition of chronic fatigue syndrome (CFS) and POTS is often found in CFS in the young. Fainting is relatively uncommon during daily life.

A major subset of POTS has increased peripheral resistance and low blood flow(LFP) related to increased angiotensin-II (Ang-II), and decreased nitric oxide (NO). NO deficits are reversed by Ang-II type-1 receptor (AT1R) blockade, ascorbic acid (AA) and tetrahydrobiopterin in skin suggesting the importance of oxidative stress. Preliminary data also suggest that the coupling of sympathetic nerve activity to blood vessel contraction is enhanced via ↑Ang-II and ↓NO. We hypothesize that this is due to activation of reactive oxygen species (ROS) including superoxide, which scavenges NO to generate peroxynitrite, and hydrogen peroxide. Combined measurements in the skin and the systemic circulation will be combined with local measurement of ROS production and sympathetic nerve activity will enable us to determine precisely how the autonomic nervous system is affected by the illness. Methods include cutaneous microdialysis to measure ROS, skin biopsy and blood tests to measure gene expression of nitric oxide synthase and Ang-II receptors, and peroneal microneurography to measure muscle sympathetic nerve activity (MSNA). Combined with ultrasonic femoral artery blood flow this will yield assessment of the interactions of nerves with the blood vessels that they control.

If we discover specific biochemical mechanisms of POTS in patients, then we may be able to specifically treat the defect.

ELIGIBILITY:
Inclusion Criteria:

* Cases will be between the ages of 14 and 29 years old referred for evaluation of orthostatic intolerance with 3 or more of the following symptoms for at least 3 months:

  * dizziness
  * nausea and vomiting
  * palpitations
  * fatigue
  * headache
  * exercise intolerance
  * blurred vision
  * abnormal sweating heat.
* Cases will have the diagnosis of symptomatic postural tachycardia made during a screening tilt table test.
* Cases will have normal physical examination, and normal electrocardiographic and echocardiographic evaluations.
* Only those free from heart disease, and from systemic illness will be eligible to participate.
* This excludes patients with illnesses and disease states known to be associated with endothelial cell dysfunction such as diabetes, renal disease, congestive heart failure, systemic hypertension, acute and chronic inflammatory diseases, neoplasm, immune mediated disease, trauma, morbid obesity and peripheral vascular disease.
* At the time of testing all patients and control subjects must refrain from vasoactive drugs for two weeks. Please check with us about any medication that you are taking.

Exclusion Criteria:

* Criteria for initial exclusion will include a condition known to be associated with endothelial dysfunction
* An active medical condition that may explain the diagnosis
* A previous medical condition with undocumented resolution that may explain the diagnosis
* Past or present major psychiatric disorder
* Substance abuse within 2 years before onset of symptoms.

Ages: 14 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2010-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Orthostatic tolerance measured by the heart rate and blood pressure response to upright tilt | 2 months

SECONDARY OUTCOMES:
Sympathetic activation and blood flow measured by sympathetic nerve recordings and Doppler blood flow in the leg | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Julian M Stewart, MD, PhD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College/Bradhurst building, Hawthorne, New York, United States

REFERENCES:
- See also: The Center for Hypotension — http://syncope.org/